CLINICAL TRIAL: NCT01783340
Title: Immunization With Plasmodium Falciparum Sporozoites Under Chloroquine or Chloroquine/Azithromycin Prophylaxis
Acronym: MMV
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: No funding
Sponsor: Radboud University Medical Center (Other)
Collaborators: Leiden University Medical Center (Other); Medicines for Malaria Venture (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MMV; NL42517.000.12 (Other: CCMO)
Record Dates: First submitted 2013-01-31; First posted 2013-02-04 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Malaria, Falciparum
Keywords: Malaria; P falciparum; Chloroquine; Azithromycin; Immunization
MeSH Terms: conditions — Malaria, Falciparum; Malaria | interventions — Azithromycin; Immunization

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- CQ and falciparum immunization (Active Comparator): This arm will receive chloroquine prophylaxis, a placebo during immunizations and three times 5 infected mosquito-bites (immunizations). Standard Chloroquine prophylactic regime: a loading dose of 300 mg on day 1 and day 3 and then 300 mg once a week, starting on day 7, for a total duration of 13 weeks.
  Placebo capsules daily on three consecutive days starting on each of three immunization days.
  Challenge: Exposure to the bites of 5 Plasmodium falciparum infected mosquitoes.
  When thick smear positive, of at day 21 after challenge, a standard 3 day treatment of Malarone will be given.
  Interventions: Drug: Placebo; Biological: Immunization with falciparum
- CQ/AZM and falciparum immunization (Experimental): This arm will receive chloroquine and azithromycin prophylaxis and three times 5 infected mosquito-bites (immunizations).
  Standard Chloroquine prophylactic regime: a loading dose of 300 mg on day 1 and day 3 and then 300 mg once a week, starting on day 7, for a total duration of 13 weeks.
  Azithromycin capsules 1000mg daily on three consecutive days starting on each of three immunization days.
  Challenge: Exposure to the bites of 5 Plasmodium falciparum infected mosquitoes.
  When thick smear positive, of at day 21 after challenge, a standard 3 day treatment of Malarone will be given.
  Interventions: Drug: Azithromycin capsules; Biological: Immunization with falciparum
- CQ and AZM control (Placebo Comparator): This arm will receive chloroquine and azithromycin prophylaxis and three times 5 uninfected mosquito-bites during immunization. Standard Chloroquine prophylactic regime: a loading dose of 300 mg on day 1 and day 3 and then 300 mg once a week, starting on day 7, for a total duration of 13 weeks.
  Azithromycin capsules 1000mg daily on three consecutive days starting on each of three immunization days.
  Challenge: Exposure to the bites of 5 Plasmodium falciparum infected mosquitoes.
  When thick smear positive, of at day 21 after challenge, a standard 3 day treatment of Malarone will be given.
  Interventions: Drug: Azithromycin capsules

INTERVENTIONS:
Drug: Azithromycin capsules — Azithromycin capsules will be administered at each immunization
  Other Names: Zithromax
  Arms: CQ and AZM control; CQ/AZM and falciparum immunization
Drug: Placebo — Placebo capsules will be administered at each immunization
  Arms: CQ and falciparum immunization
Biological: Immunization with falciparum — three inoculations with 5 infected mosquito bites
  Arms: CQ and falciparum immunization; CQ/AZM and falciparum immunization

SUMMARY:
This study will assess the superior protective immunity of the combination of chloroquine and azithromycin prophylaxis under Chemoprophylaxis Sporozoites (CPS) immunization versus a standard chloroquine prophylactic regimen.

DETAILED DESCRIPTION:
This study assesses the superiority of protective immunity of the combination of chloroquine and azithromycin prophylaxis under Chemoprophylaxis Sporozoites (CPS) immunization versus a standard chloroquine prophylactic regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤ 35 years healthy volunteers (males or females)
2. Good health based on history and clinical examination
3. Negative pregnancy serum test
4. For females who are sexually active: use of adequate contraception (incl. condom use)
5. Signing of the informed consent form, thereby demonstrating understanding of the meaning and procedures of the study
6. Agreement to inform the general practitioner and to sign a request to release medical information concerning contra-indications for participation in the study
7. Willingness to undergo a Pf controlled infection through mosquito bites
8. Agreement to stay in a hotel room close to the trial centre during a part of the study (Day 7 till day 15 after challenge)
9. Reachable (24/7) by mobile phone during the whole study period
10. Available to attend all study visits
11. Agreement to refrain from blood donation or for other purposes, during the whole study period
12. Willingness to undergo HIV, hepatitis B and hepatitis C tests
13. Negative urine toxicology screening test at screening visit and the day before challenge
14. Willingness to take a prophylactic regime of chloroquine or chloroquine/azithromycin combination and a curative regimen of Malarone® after challenge.

Exclusion Criteria:

1. History of malaria
2. Plans to travel to malaria endemic areas during the study period
3. Plans to travel outside of the Netherlands during the challenge period
4. History of stay in malaria endemic areas for more than 6 months
5. Previous participation in any malaria vaccine study and/or positive serology for Pf
6. Symptoms, physical signs and laboratory values suggestive of systemic disorders including renal, hepatic, cardiovascular, pulmonary, skin, immunodeficiency, psychiatric, and other conditions which could interfere with the interpretation of the study results or compromise the health of the volunteer
7. History of diabetes mellitus or cancer (except basal cell carcinoma of the skin)
8. History of arrhythmias or prolonged QT-interval
9. Positive family history in 1st and 2nd degree relatives for cardiac events < 50 years old
10. An estimated, ten year risk of fatal cardiovascular disease of ≥5%, as estimated by the Systematic Coronary Risk Evaluation (SCORE) system
11. Clinically significant abnormalities in electrocardiogram (ECG) at screening
12. Body Mass Index (BMI) below 18 or above 30 kg/m2
13. Any clinically significant deviation from the normal range in biochemistry or haematology blood tests or in urine analysis
14. Positive HIV, HBV or HCV tests
15. Participation in any other clinical study within 30 days prior to the onset of the study
16. Enrolment in any other clinical study during the study period
17. Pregnancy or lactation for women
18. Volunteers unable to give written informed consent
19. Volunteers unable to be closely followed for social, geographic or psychological reasons
20. History of (soft) drugs or alcohol abuse interfering with normal social function
21. A history of treatment for psychiatric disease
22. A history of epileptic insults in the volunteer
23. Contra-indications for use of Malarone®, chloroquine or azithromycin. This includes hypersensitivity or treatment taken by the volunteer that interferes with mentioned study drugs.
24. The use of chronic immunosuppressive drugs, antibiotics, or other immune modifying drugs within three months of study onset (topical corticosteroids and oral anti-histaminic are allowed) and during the study period
25. Any confirmed or suspected immunosuppressive or immunodeficient condition, including (functional) asplenia
26. Co-workers or trainees of the departments of Medical Microbiology, Parasitology, or Internal Medicine of the Leiden University Medical Centre
27. A history of sickle cell anaemia, sickle cell trait, thalassemia, thalassemia trait or G6PD deficiency

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2013-04; Primary Completion 2013-12 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Volunteers falciparum positive by thick smear | One year
  Percentage of P. falciparum thick smear negative volunteers on day 21 (protection against challenge infection)

SECONDARY OUTCOMES:
Duration of pre-patent period by thick smear | One year
  Duration of pre-patent period after challenge infection as measured by microscopy (thick smear)
Kinetics of parasitemia by PCR | One year
  Development of parasitemia as measured by PCR
Adverse events | One year
  Frequency of adverse events in study groups
Immune responses | One year
  Immune responses between study groups

CONTACTS AND LOCATIONS:
Overall Officials: RW Sauerwein, MD PhD, Study Director — Radboud University Medical Center; LG Visser, MD PhD, Principal Investigator — Leiden University Medical Centre
Locations (1):
- Leiden University Medical Centre, Leiden, Leiden, Netherlands

REFERENCES:
- [Result] Roestenberg M, McCall M, Hopman J, Wiersma J, Luty AJ, van Gemert GJ, van de Vegte-Bolmer M, van Schaijk B, Teelen K, Arens T, Spaarman L, de Mast Q, Roeffen W, Snounou G, Renia L, van der Ven A, Hermsen CC, Sauerwein R. Protection against a malaria challenge by sporozoite inoculation. N Engl J Med. 2009 Jul 30;361(5):468-77. doi: 10.1056/NEJMoa0805832. PMID 19641203